CLINICAL TRIAL: NCT02198469
Title: A Randomized, Prospective Study Comparing Methyl Aminolaevulinate Photodynamic Therapy With and Without Er:YAG Ablative Fractional Laser Treatment for Actinic Cheilitis
Brief Title: Study of Methyl Aminolaevulinate Photodynamic Therapy With and Without Er:YAG Laser in Actinic Cheilitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A University (Other)
Responsible Party: Principal Investigator, Song Ki-Hoon, Associate Professor, Dong-A University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: DAUderma-03
Record Dates: First submitted 2014-07-22; First posted 2014-07-23 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Actinic Cheilitis
Keywords: actinic cheilitis; Er:YAG ablative fractional laser; methyl aminolevulinate photodynamic therapy
MeSH Terms: conditions — Actinic cheilitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Er:YAG AFL-PDT (Experimental): Eligible patients were successively randomised to receive treatment with a single session of Er:YAG AFL MAL-PDT or 2 sessions of MAL-PDT with a 1-week interval between sessions
  Interventions: Drug: Er:YAG AFL-PDT
- MAL-PDT (Active Comparator): Eligible patients were successively randomised to receive treatment with a single session of Er:YAG AFL MAL-PDT or 2 sessions of MAL-PDT with a 1-week interval between sessions
  Interventions: Drug: MAL-PDT

INTERVENTIONS:
Drug: Er:YAG AFL-PDT — Er:YAG AFL was performed with 350 µm ablation depth, level 1 coagulation, 22% treatment density, and a single pulse. MAL cream was then applied under occlusion for 3 hrs and illuminated with a red light-emitting diode light at 37 J/cm2.
  Other Names: Er:YAG ablative fractional laser-assisted MAL-PDT
  Arms: Er:YAG AFL-PDT
Drug: MAL-PDT — a 1-mm thick layer of MAL (16% Metvix® cream, PhotoCure ASA, Oslo, Norway) was applied to the lesion and to 5 mm of surrounding healthy tissue. The area was covered with an occlusive dressing (Tegaderm, 3M, Saint Paul, MN, US) for 3 hours, after which the remaining cream was removed with saline gauze, and the red fluorescence of porphyrins was visualized with Wood's light. Each treatment area was then separately illuminated with red light-emitting diode (LED) lamps (Aktilite CL128; Galderma, Bruchsal, Germany) with peak emission at 632 nm and total light dose of 37 J cm-2. Areas scheduled to receive MAL-PDT received the second treatment 7 days later.
  Other Names: methyl aminolaevulinate-Photodynamic therapy
  Arms: MAL-PDT

SUMMARY:
Methyl aminolaevulinate photodynamic therapy (MAL-PDT) is advantageous in that it has few cosmetic side effects and minimises patient discomfort. However, its relatively low efficacy prevents its application to the treatment of actinic cheilitis(AC). Er:YAG ablative fractional laser (AFL) treatment removes the stratum corneum to increase MAL uptake and may improve efficacy. However, no studies have directly compared the efficacy of MAL-PDT with and without Er:YAG AFL in treating AC

DETAILED DESCRIPTION:
Actinic cheilitis (AC) is a keratinocytic neoplasm of the lip, especially the lower lip, is confined to the epidermis, and results from chronic or excessive ultraviolet exposure. AC is an early manifestation of lip squamous cell carcinoma (SCC), and SCC of the lip is usually associated with an identifiable pre-existent AC. Furthermore, the likelihood that AC will progress to SCC is higher than actinic keratosis (AK). Consequently, early identification and treatment of AC is recommended. PDT involves the activation of a photosensitizer by irradiation with 400- to 700-nm light to create cytotoxic oxygen and free radicals that kill dysplastic cells.

Methyl aminolaevulinate photodynamic therapy (MAL-PDT) is advantageous in that it has few cosmetic side effects and minimises patient discomfort. However, its relatively low efficacy prevents its application to the treatment of actinic cheilitis(AC).

Erbium:yttrium-aluminium-garnet (Er:YAG) ablative fractional laser (AFL) therapy has been used frequently to improve treatment efficacy of PDT. Er:YAG AFL can ablate stratum corneum with minimal penetration depth and producing minimal thermal injury. This approach creates microscopic vertical holes in the ablated tissue, surrounded by thin layers of coagulated tissue. Er:YAG AFL does not injure the entire thickness of the epidermis; therefore, healing times are minimised. Erbium:yttrium-aluminium-garnet (Er:YAG) ablative fractional laser (AFL) has been proven in recent studies to facilitate the delivery and uptake of topical MAL deep into the skin, enhancing porphyrin synthesis and photodynamic activation.

The aim of our study was to compare efficacy, recurrence rate, cosmetic outcome, and safety between Er:YAG AFL-assisted MAL-PDT (Er:YAG AFL MAL-PDT) and standard MAL-PDT in patients with AC.

ELIGIBILITY:
Inclusion Criteria:

* Korean patients ≥ 18 years of age who had biopsy-confirmed AC lesions

Exclusion Criteria:

* porphyria
* known allergies to the MAL cream or lidocaine
* pregnancy
* lactation
* any active systemic infectious disease
* immunosuppressive treatment
* personal history of malignant melanoma
* tendency towards melasma or keloid formation
* prior treatment of the lesions within 4 weeks
* any indication of poor compliance

Ages: 18 Years to 92 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Difference the efficacy between Er:YAG AFL-assisted MAL-PDT (Er:YAG AFL MAL-PDT) and standard MAL-PDT. | Efficacy was evaluated at 3 months and 12 months after treatment
  Lesion response was classified as either complete (complete disappearance of the lesion) or incomplete (incomplete disappearance) on the basis of visual examination and palpation. The response of each lesion was clinically evaluated

SECONDARY OUTCOMES:
Difference of the cosmetic outcomes between Er:YAG AFL-assisted MAL-PDT (Er:YAG AFL MAL-PDT) and standard MAL-PDT. | Cosmetic outcome was assessed by each investigator for all lesions that achieved a complete response at 12 months
  It was graded using a 4-point scale: excellent (only slight occurrence of redness or change in pigmentation), good (moderate redness or change in pigmentation), fair (slight-to-moderate scarring, atrophy, or induration), or poor (extensive scarring, atrophy, or induration)

OTHER OUTCOMES:
Difference of the recurrence rates and safety between Er:YAG AFL-assisted MAL-PDT (Er:YAG AFL MAL-PDT) and standard MAL-PDT | within 12 months after both treatment
  If the case of complete response of lesions, all patients were reviewed at 12 months to check recurrence.
  Adverse events reported by the patient were noted at each follow-up visit, including severity, duration, and need for additional therapy. All events due to PDT were described as phototoxic reactions(e.g. erythema, burning sensation, swelling, bleeding)

CONTACTS AND LOCATIONS:
Locations (1):
- Dong-A University, Busan, Dong Dae Sin-dong, Seo-gu, South Korea